CLINICAL TRIAL: NCT05715372
Title: Genetic Evaluation and Modification of Lifestyles to Improve Female Life Expectancy
Acronym: GEMLIFE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no further funding
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Barbara Soltes, MD, Professor, Department of Obstetrics and Gynecology, Rush University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 20031704
Record Dates: First submitted 2021-06-21; First posted 2023-02-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Menopause Syndrome; Inflammation; Inflammatory Response; Aging; Menopause; Telomere Shortening; Stress Oxidative
Keywords: Menopause; Inflammation; Aging; Telomeres; Oxidative Stress; Lifestyle Changes; Mindfulness; Diet; Physical Activity
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Diet, Mediterranean; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded prospective study.
Who Masked: Participant
Masking Description: Computer-assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group of menopausal women on hormone replacement (Active Comparator): This group of women on hormone replacement will have specific, structured diet, physical activity, and mindfulness-based stress reduction programs.
  Interventions: Behavioral: Mediterranean diet; Behavioral: AHA walking program; Behavioral: Mindfulness-based stress reduction
- Control group of menopausal women on hormone replacement (Placebo Comparator): This group of women on hormone replacement will be given unstructured guidelines for diet, physical activity, and stress-reduction.
  Interventions: Behavioral: Unstructured Mediterranean diet; Behavioral: Unstructured walking program; Behavioral: Unstructured stress reduction
- Intervention group of menopausal women without hormone replacement (Active Comparator): This group of women will have specific, structured diet, physical activity, and mindfulness-based stress reduction programs.
  Interventions: Behavioral: Mediterranean diet; Behavioral: AHA walking program; Behavioral: Mindfulness-based stress reduction
- Control group of menopausal women without hormone replacement (Placebo Comparator): This group of women will be given unstructured guidelines for diet, physical activity, and stress-reduction.
  Interventions: Behavioral: Unstructured Mediterranean diet; Behavioral: Unstructured walking program; Behavioral: Unstructured stress reduction

INTERVENTIONS:
Behavioral: Mediterranean diet — 12-week structured program for Mediterranean diet.
  Arms: Intervention group of menopausal women on hormone replacement; Intervention group of menopausal women without hormone replacement
Behavioral: AHA walking program — 12-week structured AHA walking program.
  Arms: Intervention group of menopausal women on hormone replacement; Intervention group of menopausal women without hormone replacement
Behavioral: Mindfulness-based stress reduction — 8-week structured mindfulness-based stress reduction (Cabot).
  Arms: Intervention group of menopausal women on hormone replacement; Intervention group of menopausal women without hormone replacement
Behavioral: Unstructured Mediterranean diet — Unstructured 12-week program with basic outline for Mediterranean diet.
  Arms: Control group of menopausal women on hormone replacement; Control group of menopausal women without hormone replacement
Behavioral: Unstructured walking program — Unstructured 12-week walking program.
  Arms: Control group of menopausal women on hormone replacement; Control group of menopausal women without hormone replacement
Behavioral: Unstructured stress reduction — Unstructured program using mobile application for stress reduction.
  Arms: Control group of menopausal women on hormone replacement; Control group of menopausal women without hormone replacement

SUMMARY:
The GEMLIFE Study is a 12-month clinical trial for menopausal women. The purpose of this study is to promote an improved aging process for women in menopause through lifestyle changes. The changes will include a heart healthy diet, structured walking program, and mindfulness-based stress reduction. During the study, the investigators will monitor components of your genetic make-up that will tell us how you are aging. Investigators will also monitor bloodwork for inflammation that can affect medical conditions. Study participants may qualify if you are within 5 years of your last menstrual period and have well controlled medical conditions. There is no cost to participants to enroll in the study- only potential benefits to the participant's health and aging process.

DETAILED DESCRIPTION:
The long-term goal of this research is to create and implement lifestyle interventions that will prevent or delay morbidities associated with accelerated aging in the menopausal women. By the end of this year, it is estimated that approximately 50 million women will be in the menopausal phase of their life. Menopause is defined by the decline in estrogen levels and subsequent increase in inflammatory markers which are associated with multiple morbidities involving the brain, bone and cardiovascular systems. Various lifestyle changes have been found to prevent or decrease these morbidities. Hormone replacement therapy in the early years of menopause is also a known therapeutic modality for the treatment of menopausal symptoms. The investigators will evaluate if hormone replacement and lifestyle change will have an enhanced effect on the prevention of morbidity and mortality.

Telomeres are distinct structures found at the end of chromosomes. As women enter into menopause, which is the biomarker for aging, there is a shortening of the telomere length. Poor lifestyle factors which cause oxidative stress, can lead to poor cell replication and critical shortening of telomere length. Telomerase, an enzyme which aids in gene sequencing, also declines. Shortened telomere length and low levels of telomerase lead to cell aging and apoptosis, a reduction in normal organ function, and an increase in morbidity and mortality. It has been found that lifestyle intervention, and possibly hormone replacement, can enhance telomere length and telomerase production.

This research will focus on the acute menopausal woman (within 5 years of the last menstrual period), with and without hormone replacement, .and multiple lifestyle interventions. Early intervention within the first five years of menopause is most important in affecting long term morbidity and mortality in women. Serial measurement of various biomarkers and cytokines associated with aging, and measurements of telomere length and telomerase levels will be performed over a 9 month period of time. Evidence shows that diet, physical activity and cognitive intervention may synergize when combined in a multimodal intervention as each targets different mechanisms. The Investigators will evaluate the efficacy of each 12-week interventions on telomere length, telomere production, serum biomarkers and cytokine levels before and after each intervention, and as a multimodal approach. Approximately 100 women will be recruited once they have been confirmed to be in the early stages of menopause, then further divided based on the use of hormone replacement. Aims are to: (1) determine the independent and combined efficacies of lifestyle interventions on telomere length, (2) determine the independent and combined efficacies of lifestyle interventions on biomarkers and and cytokines, (3) Determine other mechanisms of aging associated with the acute phase of menopause . This key knowledge will aid in practical and early lifestyle interventions to deter detrimental morbidities in the menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Non-hysterectomized women: Amenorrhea > 12 consecutive months
* Hysterectomized women: Bilateral oophorectomy (3 months after surgery)
* Normal mammogram in the past year
* Normal pap smear deemed to be negative within 5 years
* Able to understand the protocol and sign an informed consent
* Able to participate in a structured diet program for 12 weeks
* Able to participate in a structured walking program for 12 weeks
* Able to participate in a structured mindfulness-stress reduction program
* Able to operate an I-PAD, and able to connect to the internet

Exclusion Criteria:

* Known or suspected pregnancy
* Undiagnosed abnormal vaginal bleeding
* Known or suspected breast cancer or estrogen-dependent neoplasia
* Known or at risk for a MI, PE or significant cardiovascular event
* Poorly controlled blood pressure : sitting systolic > 160 or diastolic >95 mmHg
* Poorly controlled diabetes
* Uncontrolled thyroid disease
* Impaired liver function
* Unstable psychiatric disorder including depression or anxiety, PTSD
* History of drug or alcohol abuse
* Treatment with anticoagulants ( heparin, warfarin, lovenox, eliquis)
* Severe systemic disease which might interfere with interpretation of results
* Unwilling or unable to follow a diet, exercise or stress reduction protocol

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women.
Enrollment: 5 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Independent Lifestyle Interventions on Telomere Length | 12 months
  Measurement of telomere length after 12 months of a Mediterranean diet, American Heart Association walking program, and mindfulness-based stress reduction program.

SECONDARY OUTCOMES:
Lifestyle Interventions on Inflammatory Biomarkers and Cytokines | 12 months
  Inflammatory biomarkers ( C-Reactive Protein, WBC count) and cytokines (IL-6, TNFa)will be measured before 12 months of Mediterranean diet, the American Heart Association walking program and mindfulness based stress reduction
Measurement of Interventions on Inflammatory Biomarkers and Cytokines | 12 months
  Inflammatory biomarkers C-Reactive Protein, WBC count)after 12 months after a Mediterranean diet, American Heart Association walking program and mindfulness based stress reduction program

OTHER OUTCOMES:
Measurement of Menopausal aging due to stress and inflammation of the microbiome | 12 months
  Measurement of association between levels of cytokines (IL-6,TNFa)in the microbiome and telomere length

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Soltes, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Menopause study website-Gem-Life study — https://www.rushu.rush.edu
- See also: Menopause study social media page — https://www.facebook.com/GEMLIFEStudy